CLINICAL TRIAL: NCT03114280
Title: Induction Therapy With Docetaxel, Cisplatin, 5-Fluoro Uracil and Pembrolizumab in Untreated Locally-advanced Unresectable Squamous Cell Head and Neck Carcinoma (Pembrolizumab and Induction Chemotherapy in Head and Neck Squamous Cell Carcinoma. PICH Study)
Brief Title: Pembrolizumab and Induction Chemotherapy in Head and Neck Squamous Cell Carcinoma (PICH Study)
Acronym: PICH
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: MSD would not able to support the study's continuation after protocol modifications required by ANSM through dose de-escalation of pembrolizumab
Sponsor: Centre Antoine Lacassagne (Other)
Collaborators: GORTEC (Other); GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/13
Record Dates: First submitted 2017-04-02; First posted 2017-04-14 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy; Carboplatin

STUDY DESIGN:
Intervention Model Description: Fluorouracil (F) and pembrolizumab every 21 days followed by radiotherapy (RT) combined with carboplatin in untreated unresectable locally-advanced Head and Neck Squamous Cell Carcinoma (HNSCC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TPF2 (Experimental): docetaxel (T), cisplatin (P), 5 Fluorouracil (F) and pembrolizumab every 21 days followed by radiotherapy (RT) combined with carboplatin
  Interventions: Drug: TPF2; Other: Radiotherapy with carboplatin

INTERVENTIONS:
Drug: TPF2 — Combination drugs : docetaxel (T), cisplatin (P), 5 Fluorouracil (F) and pembrolizumab every 21 days
Other: Radiotherapy with carboplatin — Radiotherapy (RT) combined with carboplatin

SUMMARY:
Non-randomized phase I/II, open-labeled clinical study, 1-arm, multicenter, of docetaxel (T), cisplatin (P), 5-fluorouracil (F) and pembrolizumab every 21 days for 3 cycles followed by radiotherapy (RT) combined with carboplatin in untreated unresectable locally-advanced Head and Neck Squamous Cell Carcinoma (HNSCC).

The TPF and pembrolizumab combination will be called TP²F.

DETAILED DESCRIPTION:
The importance of intact immune surveillance in controlling outgrowth of neoplastic transformation has been known for decades. Accumulating evidence shows a correlation between tumor-infiltrating lymphocytes (TILs) in cancer tissue and favorable prognosis in various malignancies. In particular, the presence of CD8+ T-cells and the ratio of CD8+ effector T-cells / FoxP3+ regulatory T-cells seems to correlate with improved prognosis and long-term survival in many solid tumors.

The PD-1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. The normal function of PD-1, expressed on the cell surface of activated T-cells under healthy conditions, is to down-modulate unwanted or excessive immune responses, including autoimmune reactions. PD-1 (encoded by the gene Pdcd1) is an Ig superfamily member related to CD28 and CTLA-4, which has been shown to negatively regulate antigen receptor signaling upon engagement of its ligands (PD-L1 and/or PD L2). The structure of murine PD-1 has been resolved. PD-1 and family members are type I transmembrane glycoproteins containing an Ig Variable-type (V-type) domain responsible for ligand binding and a cytoplasmic tail, which is responsible for the binding of signaling molecules. The cytoplasmic tail of PD-1 contains 2 tyrosine-based signaling motifs, an immunoreceptor tyrosine-based inhibition motif (ITIM) and an immunoreceptor tyrosine-based switch motif (ITSM). Following T-cell stimulation, PD 1 recruits the tyrosine phosphatases SHP-1 and SHP-2 to the ITSM motif within its cytoplasmic tail, leading to the dephosphorylation of effector molecules such as CD3ζ, PKCθ and ZAP70 which are involved in the CD3 T-cell signaling cascade. The mechanism by which PD-1 down modulates T-cell responses is similar to, but distinct from, that of CTLA-4 as both molecules regulate an overlapping set of signaling proteins. PD-1 was shown to be expressed on activated lymphocytes including peripheral CD4+ and CD8+ T-cells, B-cells, T regs and Natural Killer cells. Expression has also been shown during thymic development on CD4-CD8- (double negative) T-cells as well as subsets of macrophages and dendritic cells. The ligands for PD-1 (PD-L1 and PD-L2) are constitutively expressed or can be induced in a variety of cell types, including non-hematopoietic cells (various tumor cells and stromal cells) as well as hematopoetic myeloid cells (dendritic cells and macrophages…). Both ligands are type I transmembrane receptors containing both IgV- and IgC-like domains in the extracellular region and contain short cytoplasmic regions with no known signaling motifs. Binding of either PD-1 ligand to PD-1 inhibits T-cell activation triggered through the T-cell receptor. PD-L1 is expressed at low levels on various non-hematopoietic tissues, most notably on vascular endothelium, whereas PD-L2 protein is only detectably expressed on antigen-presenting cells found in lymphoid tissue or chronic inflammatory environments. PD-L2 is thought to control immune T-cell activation in lymphoid organs, whereas PD-L1 serves to dampen unwarranted T-cell function in peripheral tissues. Although healthy organs express little (if any) PD-L1, a variety of cancers were demonstrated to express abundant levels of this T-cell inhibitor. PD-1 has been suggested to regulate tumor-specific T-cell expansion in subjects with melanoma (MEL). This suggests that the PD-1/PD-L1 pathway plays a critical role in tumor immune evasion and should be considered as an attractive target for therapeutic intervention.

Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. KeytrudaTM (pembrolizumab) has recently been approved in the United Stated for the treatment of patients with unresectable or metastatic melanoma and disease progression following ipilumumab and, if BRAF V600 mutation positive, a BRAF inhibitor.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in this trial, the subject should fulfill the following criteria:

1. Age > or = 18 and < 70 years years at the time of signing informed consent,
2. Histologically or cytologically confirmed head and neck squamous-cell carcinoma (oral cavity, oropharynx and hypopharynx) with locoregionally-advanced disease stage III or IV without metastasis, previously untreated,
3. Measurable disease based on RECIST 1.1,
4. Performance status of 0 or 1 on the ECOG Performance Scale,
5. Adequate organ function described in protocol section 4.2 - Inclusion criteria,
6. Tumors considered unresectable by a multidisciplinary team,
7. Available biopsy sample and HPV status,
8. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required,
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 180 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year,
10. Male subjects should agree to use an adequate method of contraception or abstain from heterosexual activity starting with the first dose of study therapy through 180 days after the last dose of study therapy,
11. Patient willing and able to provide written informed consent/assent for the trial,
12. Patient affiliated with a health insurance system.

Exclusion criteria

The subject should not enter into the study if any of the following exclusion criteria are fulfilled:

1. Tumors of the nasopharynx, larynx and the nasal and paranasal cavities,
2. Hemorrhagic tumors, Protocol PICH_version 2.0 of 02 May 2018 Page 10 sur 127
3. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of treatment,
4. Before the first dose of trial treatment:

   a) Had major surgery (< 4 weeks prior to the first dose), Note: If subject received major surgery, he must have recovered adequately from the toxicity and/or complications from the intervention before starting therapy,
5. Diagnosis of immunodeficiency (including HIV 1/2 positivity) or currently received systemic steroid therapy with dose superior to 10 mg/day of prednisone or equivalent or any other form of immunosuppressive therapy, within 7 days prior to the first dose of trial treatment,
6. Known history of active Bacillus Tuberculosis (TB),
7. Hypersensitivity to pembrolizumab or any of its excipients,
8. Any contraindication for receiving a treatment of docetaxel, cisplatin, 5-fluorouracil or carboplatin,
9. Hearing impairment or cardiorespiratory pathology with a contraindication of overhydration,
10. Currently received prophylactic treatment of phenytoin which could have an interaction with cisplatin, 5-fluorouracile or carboplatin or fosphenytoin which could have an interaction with carboplatin,
11. Currently received treatment of sorivudine or analogues (e.g. brivudine) with could have an interaction with 5-fluorouracile,
12. Complete known dihydropyrimidine dehydrogenase deficiency (DPD),
13. Clinically active cardiac disease or myocardial infarction within 6 months prior to the first dose of treatment,
14. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer,
15. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc…) is not considered a form of systemic treatment,
16. History of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis,
17. Active infection requiring systemic therapy,
18. History or current evidence of any condition, therapy, or laboratory abnormality that might influence the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator,
19. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial,
20. Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the pre-screening or screening visit through 180 days after the last dose of trial treatment,
21. Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent,
22. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected),
23. Received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed. However, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed,
24. Received prior organ transplant which may include an allogenic stem cell transplant,
25. People particularly vulnerable as defined in Articles L.1121-5 to -8 of the French Healthcare Code, including: person deprived of freedom by an administrative or judicial decision, adult being the object of a legal protection measure or outside a state to express their consent, pregnant or breastfeeding women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Phase I : Evaluation of Recommended dose for phase II and characterization of the safety and tolerability profile of pembrolizumab when administered in combination with docetaxel, cisplatin and 5 Fluorouracil | 12 months post treatment
  To evaluate by using a "3+3 modified schedule" the Recommended Phase 2 Dose (RPD2), Dose Limiting Toxicities (DLT) and Maximal Tolerated Dose (MTD) of the association of pembrolizumab with induction therapy by docetaxel, cisplatin and 5-fluorouracil (TP²F) as first-line treatment for patients with locally-advanced unresectable HNSCC
Phase II : Progression-free survival | 12 months post treatment
  Progression-free survival : To evaluate, in terms of progression-free survival rate at 12 months, the efficacy of the association of pembrolizumab with induction therapy by docetaxel, cisplatin and 5-fluorouracil (TP²F) as first-line treatment for patients with locally-advanced unresectable HNSCC ; in order to demonstrate that the addition of pembrolizumab to TPF can increase efficacy without increasing toxicity.

SECONDARY OUTCOMES:
Phase I : Antitumor activity | 24 months post treatment
  To document any antitumor activity observed with pembrolizumab in combination with docetaxel, cisplatin and 5 Fluorouracil
Phase II : Overall survival rate | 24 months post treatment
  Overall survival rate at 2 years. It will be calculated from the date of study inclusion to the date of the event or to the last known contact of the patient, for those still event free at the time of the last follow-up until 24 months post treatment.
Phase II : Best Overall response | 24 months post treatment
  Best overall response rate after induction chemotherapy : Partial Response or Complete Response or Stable Disease after induction chemotherapy (qualitative data)
Phase II : Best Overall response | 24 months post treatment
  Best overall response rate after radiation therapy: Partial Response or Complete Response or Stable Disease after radiation therapy (qualitative data)
Phase II : Objective response rate | 24 months post treatment
  Objective response rate (ORR) will be determinated by evaluation of Complete Response (CR) and Partial Response (PR)
Phase II : Progression-free survival (PFS) at 12 months | 12 months
  Progression-free survival (PFS) is defined by disease recurrence. It will be calculated from the date of study inclusion to the date of the event or to the last known contact of the patient, for those still event free at the time of the last follow-up until 12 months after the treatment.
Phase II : Level of expression of PD1 before and after treatment | 7 weeks
  Level of expression of PD1 will be determinated by using quantitative and qualitative data before and after treatment
Phase II : Evaluation of Safety | 24 months
  Toxicity will be evaluated according to NCI-CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Chrisine LOVERA, Study Director — Centre Antoine Lacassagne
Locations (1):
- PEYRADE Frédéric, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided